CLINICAL TRIAL: NCT05774873
Title: A Phase I/II Study of IBI334 in Subjects With Unresectable, Locally Advanced or Metastatic Solid Tumors
Brief Title: The Primary Objective of This Study to Evaluate the Safety and Tolerability of IBI334 and Determine the Maximum Tolerated Dose (MTD) and the Recommended Phase 2 Dose (RP2D)and Anti Tumor Activity of IBI334.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI334A101
Record Dates: First submitted 2023-02-08; First posted 2023-03-20 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI334 in advanced solid tumors (Experimental)
  Interventions: Drug: IBI334

INTERVENTIONS:
Drug: IBI334 — There are six dose of IBI334 ,QW IV in first cycle and Q2W IV behind the first cycle

SUMMARY:
This is open-label, multicenter, Phase I/II study is designed to evaluate the Safety and tolerability and Efficacy of IBI334 Monotherapy in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria：

1. Subjects with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol;
2. Male or female subjects ≥ 18 years old;
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1;
4. Anticipated life expectancy of ≥ 12 weeks;
5. At least 1 evaluable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1with Phase Ia ;At least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 with Phase Ib+II；

Exclusion Criteria：

1. Participate in any other interventional clinical research except observational (non-interventional) study or in the follow-up phase of the interventional study;
2. Received live vaccines within 4 weeks prior to first dose of the study drug or plan on receiving any live vaccine during the study;
3. History of immunodeficiency disease, including congenital or acquired immunodeficiency diseases;
4. Severe allergic or hypersensitive to other EGFR or B7H3 antibodies or any ingredients of IBI334;
5. Plan to receive other antitumor therapy during the study excluding palliative radiotherapy for the purpose of symptom (like pain) relief, which must not affect tumor assessment throughout the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse events | Up to 60 days post last dose
Percentage of subjects woth Dose-Limitine toxicities(DLTs) | Up to 28 days following first dose

SECONDARY OUTCOMES:
PK profile: major PK parameters of single and multiple doses of drugs, including but not limited to: area under the curve (AUC) | Day 1 up to treatment duration reaches 24 months
PK profile: major PK parameters of single and multiple doses of drugs, including but not limited to:maximum concentration (Cmax) | Day 1 up to treatment duration reaches 24 months
PK profile: major PK parameters of single and multiple doses of drugs, including but not limited to: clearance (CL) | Day 1 up to treatment duration reaches 24 months
PK profile: major PK parameters of single and multiple doses of drugs, including but not limited to: apparent volume of distribution (V) | Day 1 up to treatment duration reaches 24 months
PK profile: major PK parameters of single and multiple doses of drugs, including but not limited to: half-life (t1/2). | Day 1 up to treatment duration reaches 24 months
Prevalence and incidence of anti-IBI334 antibodies. | Day 1 up to treatment duration reaches 24 months
Preliminary efficacy ： objective response rate (ORR) as evaluated per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria | Day 1 up to treatment duration reaches 24 months
Preliminary efficacy : duration of response (DoR) as evaluated per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria | Day 1 up to treatment duration reaches 24 months
Preliminary efficacy : disease control rate (DCR) as evaluated per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria | Day 1 up to treatment duration reaches 24 months
Preliminary efficacy :time to response (TTR) as evaluated per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria | Day 1 up to treatment duration reaches 24 months
Preliminary efficacy :progression-free survival (PFS) as evaluated per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria | Day 1 up to treatment duration reaches 24 months
Preliminary efficacy :overall survival (OS) | Day 1 up to treatment duration reaches 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Shandong First Medical university, Jinan, Shandong, China